CLINICAL TRIAL: NCT01919125
Title: A Phase I, Open-Label, Single-Dose Study to Evaluate the Pharmacokinetics of IDX719 in Subjects With Normal and Impaired Hepatic Function
Brief Title: Pharmacokinetics of IDX719 in Participants With Normal and Impaired Hepatic Function (MK-1894-008)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1894-008; IDX-06A -008
Record Dates: First submitted 2013-08-06; First posted 2013-08-08 (Estimated); Last update posted 2016-01-26 (Estimated); Status verified 2016-01

CONDITIONS: Hepatitis C, Chronic
Keywords: Chronic hepatitis C; Hepatitis C virus; HCV
MeSH Terms: conditions — Hepatitis C, Chronic; Hepatitis C | interventions — samatasvir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Cohort 1: Child-Pugh Class A (Experimental): Participants with mild hepatic impairment (Child-Pugh Class A score = 5-6) will receive a single dose of 100 mg IDX719 by mouth on Day 1.
  Interventions: Drug: IDX719
- Cohort 2: Child-Pugh Class B (Experimental): Participants with moderate hepatic impairment (Child-Pugh Class B score = 7-9) will receive a single dose of 100 mg IDX719 by mouth on Day 1.
  Interventions: Drug: IDX719
- Cohort 3: Child-Pugh Class C (Experimental): Participants with severe hepatic impairment (Child-Pugh Class C score = 10-15) will receive a single dose of 100 mg IDX719 by mouth on Day 1.
  Interventions: Drug: IDX719

INTERVENTIONS:
Drug: IDX719 — IDX719 supplied as 50 mg tablets.
  Other Names: Samatasvir

SUMMARY:
The purpose of this study is to evaluate the pharmacokinetics (PK) and safety and tolerability of single-dose administration of IDX719 in participants with normal hepatic function and participants with varying degrees of hepatic impairment.

ELIGIBILITY:
Inclusion Criteria:

* Read and sign the written informed consent form (ICF) after the nature of the study has been fully explained.
* All subjects of childbearing potential must have agreed to use a double method of birth control (one of which must be a barrier) from Screening through at least 90 days after the last dose of the study drug.
* Male subjects have agreed not to donate sperm from Day -1 through 90 days after the last dose of study drug.

Exclusion Criteria:

* Pregnant or breastfeeding.
* Other clinically significant medical conditions or laboratory abnormalities

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2013-08; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Maximum plasma concentration (Cmax) | Up to 6 days
Time to maximum plasma concentration (Tmax) | Up to 6 days
Area under the curve (AUC) from time zero to last measurable concentration (AUC0-last) | Up to 6 days
AUC from time zero to infinity (AUC0-~) | Up to 6 days
AUC from time zero to 24 hours (AUC0-24h) | Up to 6 days
Plasma concentration 24 hours after dosing (C24h) | Up to 6 days
Apparent terminal elimination rate constant | Up to 6 days
Observed terminal half-life (T1/2) | Up to 6 days

SECONDARY OUTCOMES:
Percentage of participants experiencing serious adverse events (SAEs) | Up to 6 days
Percentage of participants experiencing an adverse event (AE) | Up to 6 days
Percentage of participants experiencing Grade 1-4 laboratory abnormalities | Up to 6 days

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC